CLINICAL TRIAL: NCT07050719
Title: Can Atelectasis be Prevented in Robotic Surgery by Monitoring With Oxygen Reserve Index (ORI)? A Randomized Controlled Trial
Brief Title: Can Atelectasis Be Prevented With Oxygen Reserve Index (ORI) Monitoring?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Antalya Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Nilgun Kavrut Ozturk, PROFESSOR MD, Antalya Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: AEAHAE001
Record Dates: First submitted 2025-06-22; First posted 2025-07-03 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Atelectasis; Lung Ultrasonography Score; Hyperoxia
Keywords: Atelectasis; ORI; robotic surgery; lung ultrasound score; hyperoxia
MeSH Terms: conditions — Pulmonary Atelectasis; Hyperoxia | interventions — Oxygen Saturation; Lactoperoxidase; Population Groups

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peripheral Oxygen Saturation (SpO₂) Group (Active Comparator): FiO₂ adjusted based on pulse oximetry to maintain SpO₂ ≥98%
  Interventions: Procedure: Peripheral Oxygen Saturation (SpO₂) Group
- Peripheral Oxygen Saturation and Oxygen Reserve Index (SpO₂-ORI) Group (Active Comparator): FiO₂ adjusted using both SpO₂ and ORI to maintain ORI between 0-0.3
  Interventions: Procedure: Peripheral Oxygen Saturation and Oxygen Reserve Index (SpO₂-ORI) Group

INTERVENTIONS:
Procedure: Peripheral Oxygen Saturation (SpO₂) Group — FiO₂ adjusted based on pulse oximetry to maintain SpO₂ ≥98%
  Arms: Peripheral Oxygen Saturation (SpO₂) Group
Procedure: Peripheral Oxygen Saturation and Oxygen Reserve Index (SpO₂-ORI) Group — FiO₂ adjusted using both SpO₂ and ORI to maintain ORI between 0-0.3
  Arms: Peripheral Oxygen Saturation and Oxygen Reserve Index (SpO₂-ORI) Group

SUMMARY:
This single-center randomized controlled trial aims to evaluate whether intraoperative monitoring using the Oxygen Reserve Index (ORI) reduces the incidence of postoperative atelectasis, as assessed by lung ultrasound (LUS), in adult patients undergoing elective robotic surgery under general anesthesia.

DETAILED DESCRIPTION:
Postoperative atelectasis is observed in 60-90% of patients undergoing general anesthesia. Factors such as high inspired oxygen concentration, muscle relaxation, and reduced functional residual capacity contribute to its development through mechanisms like absorption atelectasis. The persistence of atelectasis increases the risk of pneumonia, hypoxia, prolonged hospital stay, healthcare costs, and mortality. Despite the well-known pathophysiology, the optimal intraoperative fraction of inspired oxygen (FiO₂) remains unclear.

The Oxygen Reserve Index (ORI) is a non-invasive, continuous parameter that reflects the oxygen reserve within the moderate hyperoxia range (100-200 mmHg). It may facilitate individualized FiO₂ titration to avoid hyperoxia-related atelectasis. Lung ultrasound (LUS) is a reliable, radiation-free bedside tool for detecting atelectasis.

This study hypothesizes that ORI-guided oxygen therapy will reduce the incidence of postoperative atelectasis compared to standard Peripheral Capillary Oxygen Saturation (SpO₂)-guided therapy.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists Physical Status Classification System (ASA) physical status I-III
* Elective robotic surgery under general anesthesia
* Surgery duration >2 hours
* Requires invasive arterial cannulation
* Signed informed consent

Exclusion Criteria:

* ASA IV or higher
* Room air SpO₂ <92%
* Chronic pulmonary disease
* Hemoglobinopathy
* Pregnancy
* Refusal to participate

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2025-07-15 (Actual); Primary Completion 2025-12-08 (Actual); Study Completion 2025-12-08 (Actual)

PRIMARY OUTCOMES:
Postoperative LUS score at 30 min | At 30 minutes following tracheal extubation at the end of surgery
  Lung ultrasound (LUS) measurements will be performed by an anesthesiologist blinded to the study groups, who is experienced in lung ultrasonography with at least 100 prior examinations. LUS will be performed and recorded 30 minutes before surgery while patients are in the supine position, using a linear probe (6-12 MHz). The total LUS score will be calculated as the sum of the scores for the 12 quadrants of each hemithorax (range: 0-36). Higher scores will indicate more severe loss of aeration. Loss of aeration will be scored as follows:
  * 0: Presence of A-lines or fewer than two B-lines
  * 1: Three or more well-defined B-lines
  * 2: Presence of multiple coalescent B-lines
  * 3: Presence of lung consolidation characterized by dynamic air bronchograms

SECONDARY OUTCOMES:
Preoperative LUS score | 30 minutes prior to patient transfer to the operating room
  Lung ultrasound (LUS) measurements will be performed by an anesthesiologist blinded to the study groups, who is experienced in lung ultrasonography with at least 100 prior examinations. LUS will be performed and recorded 30 minutes before surgery while patients are in the supine position, using a linear probe (6-12 MHz). The total LUS score will be calculated as the sum of the scores for the 12 quadrants of each hemithorax (range: 0-36). Higher scores will indicate more severe loss of aeration. Loss of aeration will be scored as follows: • 0: Presence of A-lines or fewer than two B-lines • 1: Three or more well-defined B-lines • 2: Presence of multiple coalescent B-lines • 3: Presence of lung consolidation characterized by dynamic air bronchograms
Intraoperative arterial partial pressure of oxygen (PaO₂) | At baseline (immediately before incision), and at 1st, 2nd, and 3rd hour intraoperatively
  Arterial blood samples will be collected intraoperatively at baseline (immediately before skin incision) and at the 1st, 2nd, and 3rd hour to measure the partial pressure of oxygen (PaO₂).
Intraoperative fraction of inspired oxygen (FiO₂) | At baseline (immediately before incision), and at 1st, 2nd, and 3rd hour intraoperatively
  The fraction of inspired oxygen administered to the patient will be recorded at baseline (immediately before skin incision) and hourly at the 1st, 2nd, and 3rd hour during surgery.
Intraoperative Oxygen Reserve Index (ORI) | At baseline (immediately before incision), and at 1st, 2nd, and 3rd hour intraoperatively
  Continuous monitoring of the Oxygen Reserve Index (ORI) will be performed, and values will be documented at baseline (immediately before skin incision) and at 1st, 2nd, and 3rd hour intraoperatively.Intraoperative Oxygen Reserve Index (ORI) will be measured. ORI is a unitless index ranging from 0.00 to 1.00, with higher values indicating a greater oxygen reserve.
Number of episodes with severe hyperoxia (PaO₂ > 200 mmHg) | At baseline (immediately before incision), and at 1st, 2nd, and 3rd hour intraoperatively
  The number of severe hyperoxia episodes, defined as PaO₂ levels exceeding 200 mmHg, will be recorded at baseline (immediately before skin incision) and at the 1st, 2nd, and 3rd hour during surgery.Each time point will be evaluated independently, and the number of measurements exceeding 200 mmHg will be counted.This is a binary threshold-based event count, not a continuous scale; thus, no scoring system or scale interpretation is applicable.

CONTACTS AND LOCATIONS:
Overall Officials: NILGUN KAVRUT OZTURK, PROFESSOR MD, Study Chair — Antalya Training and Research Hospital; AYSE MERVE ERDEM, RESIDENT, Principal Investigator — Antalya Training and Research Hospital
Locations (1):
- Antalya Training and Research Hospital, Antalya, Muratpasa, Turkey (Türkiye)